CLINICAL TRIAL: NCT05896267
Title: SpO2 Data Collection in Pediatric Patients Using INVSENSOR00061
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BAIL0003
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Spo2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Masimo INVSENSOR00061 (Experimental): Experimental: INVSENSOR00061 All subjects are enrolled into this arm will have noninvasive blood oxygen measurements obtained.
  Interventions: Device: Masimo INVSENSOR00061

INTERVENTIONS:
Device: Masimo INVSENSOR00061 — Masimo INVSENSOR00061 will be used to measure noninvasive SpO2 (Oxygen Saturation )

SUMMARY:
This is a prospective, non-randomized data collection study to evaluate the form, fit, and function of INVSENSOR00061.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is a full-term newborn (37 weeks) to 18 months of age.

Exclusion Criteria:

* • Subject has underdeveloped skin.

  * Subject has a skin condition and/or deformity at the planned application site, which would preclude sensor placement and measurements.
  * Subject has an absence or deformities of limbs or severe edema, which would interfere with sensor application or prevent the proper fit of the sensors.
  * Subject is not suitable for the investigation at the discretion of the Investigator.

Ages: 37 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bailony Pediatrics, National City, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Masimo INVSENSOR00061
Started | 64
Completed | 60
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Masimo INVSENSOR00061
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 14
  White | 38
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Accuracy of INVSENSOR00061
Description: SpO2 accuracy will be determined by calculating the Arithmetic Root Mean Square (ARMs) value which will be reported as percent of oxygen saturated hemoglobin. The noninvasive oxygen saturation measurement (SpO2) from the INVSENSOR00061 will be compared to the noninvasive oxygen saturation measurement (SpO2) value from the RD SET Neo sensor.
Time Frame: Approximately 15 minutes
Population: 30 subjects were excluded from the analysis and replaced with new participants because of incorrect sensor placement.
Measure: Number; unit: percent of oxygen saturated hemoglobin
Groups:
- Masimo INVSENSOR00061: Experimental: INVSENSOR00061 All subjects are enrolled into this arm will have noninvasive blood oxygen measurements obtained.
  Masimo INVSENSOR00061: Masimo INVSENSOR00061 will be used to measure noninvasive SpO2 (Oxygen Saturation ) in blood .
Arm/Group | Masimo INVSENSOR00061
Number analyzed (Participants) | 30
percent of oxygen saturated hemoglobin | 0.87

2. Primary Outcome: Pulse Rate Accuracy of INVSENSOR00061
Description: Pulse Rate accuracy will be determined by calculating the Arithmetic Root Mean Square (ARMs) value through the comparison of the noninvasive Pulse Rate to the noninvasive Pulse Rate (PR) value obtained from the RD SET Neo sensor which will be reported as beats per minute.
Time Frame: Approximately 15 minutes
Population: 30 subjects were excluded from the analysis and replaced with new participants because of incorrect sensor placement.
Measure: Number; unit: beats per minute
Arm/Group | Masimo INVSENSOR00061
Number analyzed (Participants) | 30
beats per minute | 4.45

ADVERSE EVENTS:
Time Frame: Approximately 30 minutes
Arm/Group | Masimo INVSENSOR00061
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT05896267/Prot_SAP_000.pdf